CLINICAL TRIAL: NCT01220791
Title: Methylprednisolone vs. Placebo to Control Late Follicular Progesterone Elevation in GnRH-Antagonist IVF Cycles
Brief Title: Methylprednisolone Addition in IVF Treatment of Infertile Couples
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Collaborators: BioGenesis (Industry); HRG (Unknown)
Responsible Party: Papanikolaou Evangelos, HRG
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Medrol005
Record Dates: First submitted 2010-08-27; First posted 2010-10-14 (Estimated); Last update posted 2010-10-14 (Estimated); Status verified 2010-10

CONDITIONS: In Vitro Fertilization
Keywords: methylprednisolone; IVF; progesterone; corticosteroid; late follicular phase; pregnancy rates
MeSH Terms: interventions — Pregnancy; Methylprednisolone; Progesterone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Follicular Medrol (Active Comparator): In an Antagonist protocol for IVF patients will also receive 4mg tabl. Methylprednisolone twice a day from the day 2 of ovarian stimulation and until the day of the pregnancy test on luteal day-14 post oocyte retrieval
  Interventions: Other: In vitro fertilization treatment for infertility
- No medrol group (Placebo Comparator): Patients will receive only Antagonist protocol for IVF as usual
  Interventions: Other: In vitro fertilization treatment for infertility

INTERVENTIONS:
Other: In vitro fertilization treatment for infertility — IVF treatment
  Other Names: pregnancy; MEDROL; progesterone

SUMMARY:
Hypothesis to be tested is whether follicular addition of Methylprednisolone can efficiently control late follicular progesterone rise during IVF treatment

DETAILED DESCRIPTION:
The aim is to investigate any potential advantages of adding cortisone supplementation from the follicular phase onwards with regard to premature luteinization, oocyte quality, embryo quality and pregnancy outcome.

ELIGIBILITY:
Inclusion Criteria:

* less than 36, more than 10 antral follicles, FSH<12

Exclusion Criteria:

* endometriosis stage III&IV,

Ages: 21 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Progesterone rise above 1.5ng.ml on the day of HCG | up to 14 days of follicular ovarian stimulation
  Incidence or high progesterone on the day of HCG triggering

SECONDARY OUTCOMES:
Clinical pregnancy rate | Follow pregnancy until delivery
  Success rate in IVF cycles

CONTACTS AND LOCATIONS:
Overall Officials: Basil Tarlatzis, Professor, Study Chair — BioGenesis
Locations (1):
- Biogenesis, Thessaloniki, Pylaia, Greece

REFERENCES:
- [Background] Bider D, Menashe Y, Goldenberg M, Dulitzky M, Lifshitz A, Dor J. Dexamethasone as an adjuvant therapy for anovulatory, normoandrogenic patients during ovulation induction with exogenous gonadotropins. J Assist Reprod Genet. 1996 Sep;13(8):613-6. doi: 10.1007/BF02069638. PMID 8897119
- See also: web page of investigator centre — http://www.hrg.gr